CLINICAL TRIAL: NCT04856241
Title: Prep-to-Play: Comparing the Impact of Supported and Unsupported Implementation Strategies on the Use of an Injury Prevention Program in Women's/Girl's Community Football
Brief Title: Making Football Safer for Women: Implementing an Injury Prevention Program
Acronym: Prep-to-Play
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: La Trobe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: P2P NHMRC 1193733
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-07

CONDITIONS: Anterior Cruciate Ligament Injuries; Concussion, Brain; Musculoskeletal Injury
Keywords: injury prevention; implementation; football; female
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Brain Concussion

STUDY DESIGN:
Intervention Model Description: Stepped-wedge randomised controlled trial. Prior to study initiation, the leagues will be randomly allocated to one of the five wedges for time of crossover from the control to the intervention phase using a computer-generated list of random numbers provided by a statistician. The randomisation sequence will be concealed to the coaches until shortly before the switch (~four weeks to allow time to organise their workshop).
Who Masked: Outcomes Assessor
Masking Description: It will not be possible to blind all involved research fellows, or the Prep-to-Play Physiotherapists involved in the project. The statistician will be unblinded to information required to complete the analyses (i.e. timing of transition) but blinded to team information (e.g. location, name). Teams will be given a unique code.
  To optimise allocation concealment: i) each cluster will be a league or leagues in a unique geographical area; ii) data collection at all sites will commence in the control period, iii) team designate and/or sports trainers will remain blinded to allocation sequence; iv) Prep-to-Play observers validating the primary outcome (Prep-to-Play implementation) will be independent to the club and blinded to allocation; v) research fellows collecting injury data will be independent of the club and blinded to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supported Implementation (Intervention) (Experimental): Our supported implementation approach is designed to improve uptake of Prep-to-Play. The Prep-to-Play program consists of four components: dynamic warm-up, strength training, football fundamentals, and education. At the start of the intervention period, Prep-to-Play Physiotherapists will conduct a 3-hour workshop for coaches and influential players. Ongoing support will be provided via a range of strategies. Prep-to-Play Physiotherapists will attend training (two times) during and immediately post implementation to provide coaches with support (feedback on missing components, player technique, questions). Monthly Coaches Shed; Online drop-in session with education component to meet other coaches (peer support & networking) and ask questions. Refresher workshops will be run in pre-season 2022 for the teams who have received the intervention in 2021.
  Interventions: Other: Coaching; Other: Peer support; Other: Educational materials
- Unsupported implementation (Control) (Active Comparator): The unsupported implementation arm will be "usual care". Access to the Prep-to-Play resources, including videos, downloadable manuals and posters, are freely available to coaches online. The online resources incorporate the same four concepts as described in the supported implementation - dynamic warm-up, strength exercises, football fundamentals, and education. In the control arm, no additional resources, education, or support will be provided.
  Interventions: Other: Educational materials

INTERVENTIONS:
Other: Coaching — Physiotherapists (trained by the research team) train the coaches to deliver Prep-to-Play. The Physiotherapists will also provide face-to-face one-to-one support to each coach at their team's training session (two visits), with all their players.
  Arms: Supported Implementation (Intervention)
Other: Peer support — Coaches shed. Coaches provide each other with support and ideas. Strategies to overcome barriers and motivate players.
  Arms: Supported Implementation (Intervention)
Other: Educational materials — Prep-to-Play program resources are available online for coaches and players to view

SUMMARY:
The aim of this study is to determine how we can best support coaches to implement an injury prevention (IP) program (Prep-to-Play) in female community Australian Football. We will recruit at least 140 female community football teams from 15 different football leagues in Victoria, Australia. Teams will be competing in U16, U17, U18, U19 or open womens competitions. We will train and support coaches to implement the IP program and evaluate the effects of the IP program on injuries across two football seasons.

DETAILED DESCRIPTION:
Primary Aim: To compare the impact of supported and unsupported implementation strategies on the use of an IP program (Prep-to-Play) in female community Australian Football.

Secondary aims are to:

1. Evaluate the effects of supported implementation of Prep-to-Play on injury risk reduction.
2. Identify barriers and enablers to sustainability of the Prep-to-Play implementation model, and develop clear recommendations for a future, sustainable national roll out of Prep-to-Play.
3. Evaluate the cost-effectiveness of Prep-to-Play.

Primary hypothesis

The primary hypothesis is that supported implementation will result in increased use of Prep-to-Play in female community Australian Football compared to unsupported implementation.

Secondary hypotheses

The secondary hypotheses are that the supported implementation of Prep-to-Play will:

* result in a reduction of anterior cruciate ligament (ACL) injuries in females participating in community Australian Football;
* result in a reduction of other musculoskeletal injuries and concussion among females participating in community Australian Football;
* be more cost-effective than the unsupported implementation.

ELIGIBILITY:
Inclusion Criteria

* Coach consents to be trained and to implement Prep-to-Play
* Team includes players aged 13 years and above registered to play community football
* The team trains at least once per week in addition to match-play
* Coach has at least Level I coach accreditation (or enrolled to be accredited in 2021)

Exclusion Criteria:

* Inability to understand written English
* Players aged less than 13 years

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 2600 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2025-04-13 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Use of Prep-to-Play (Primary outcome) | 18 months
  Use of Prep-to-Play will be calculated as the proportion of all possible team sessions (training and games) where Prep-to-Play essential components were completed.
  The primary outcome assessor will be the Team Designate (i.e., nominated team manager, or team representative) who will record (via the Smartabase App or website) whether essential components of Prep-to-Play were completed at each training session and games.
  In addition to the Team Designate, Prep-to-Play Observers (research assistants blinded to randomisation) will make five random visits (≥one prior to the intervention period and ≥two after the intervention period) to observe the execution of Prep-to-Play in order to validate team use data from the Team Designates.

SECONDARY OUTCOMES:
Number of players with an ACL injury (Secondary outcome) | 18 months
  The primary injuries of interest are ACL injuries and concussion. An ACL/all other injuries will be defined as any injury occurring during a football match or training that results in a player being unable to return to the field of play for that match, or missing at least one match.
  ACL injury definition
  • Ruptured ACL is confirmed by clinical examination, with or without magnetic resonance imaging or surgery.
  Injury data will be collected via two methods to minimise missing data: (i) sports trainer; (ii) direct from player
Number of players with a concussion (Secondary outcome) | 18 months
  A head injury will be defined as any injury to the head region occurring during a football match or training, regardless of time loss.
  Concussion definition
  • Direct or indirect impact to the head resulting in loss of consciousness and/or any of the following clinical symptoms (memory loss, headache, dizziness, nausea, difficulty concentrating, feeling like being in a fog, feeling not quite right).
  Injury data will be collected via two methods to minimise missing data: (i) sports trainer; (ii) direct from player
Number of player hours (training and match) | 18 months
  The number of training and match hours for each team will be collected, and reported at a team-level. Weekly team match exposure will be estimated from the number of matches played, multiplied by the number of players in each match (publicly available registry), and the match length (junior: 1 hour, senior: 1.5 hours). Weekly team training exposure will be estimated using the number and duration of football training sessions completed (reported by team designates), multiplied by the average number of players at training (reported by independent observers on five occasions).
Healthcare utilisation | 18 months
  Healthcare use for players sustaining a knee or head injury will be obtained by the blinded research officer to estimate healthcare costs of sustaining an injury to inform health economic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Kay Crossley, PhD, PT, Principal Investigator — La Trobe University
Locations (1):
- Community Australian Football Leagues, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patterson BE, Donaldson A, Cowan SM, King MG, Barton CG, McPhail SM, Hagglund M, White NM, Lannin NA, Ackerman IN, Dowsey MM, Hemming K, Makdissi M, Culvenor AG, Mosler AB, Bruder AM, Choong J, Livingstone N, Elliott RK, Nikolic A, Fitzpatrick J, Crain J, Haberfield MJ, Roughead EA, Birch E, Lampard SJ, Bonello C, Chilman KL, Crossley KM. Evaluation of an injury prevention programme (Prep-to-Play) in women and girls playing Australian Football: design of a pragmatic, type III, hybrid implementation-effectiveness, stepped-wedge, cluster randomised controlled trial. BMJ Open. 2022 Sep 14;12(9):e062483. doi: 10.1136/bmjopen-2022-062483. PMID 36104145